CLINICAL TRIAL: NCT02111863
Title: A Phase II Study of Cell Transfer Therapy for Metastatic Melanoma Using 41BB Selected Tumor Infiltrating Lymphocytes Plus IL-2 Following a Non-Myeloablative Lymphocyte Depleting Chemotherapy Regimen
Brief Title: Immunotherapy Using 41BB Selected Tumor Infiltrating Lymphocytes for Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to low accrual and change in research focus.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140062; 14-C-0062
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Melanoma; Skin Cancer
Keywords: Skin Cancer; Metastatic Melanoma; Adoptive Cell Therapy; Immunotherapy; Clinical Response
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — aldesleukin; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lymphocyte Depleting Prep Regimen (Experimental): Patients will receive a lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine followed by intravenous (IV) infusion of 4-1BB selected tumor infiltrating lymphocytes (TIL) plus IV aldesleukin.
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: 4-1BB Selected Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes approximately every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
  Other Names: Proleukin
Drug: Fludarabine — Fludarabine 25 mg/m^2/day (intravenous piggyback) IVPB daily X 5 days.(The fludarabine will be started approximately 1-2 hours after the cyclophosphamide on Days -5 and -4)
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml 5% dextrose in water (D5W) over 1 hr.
  Other Names: Cytoxan
Biological: 4-1BB Selected Tumor Infiltrating Lymphocytes (TIL) — On day 0, cells will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes (one to four days after the last dose of fludarabine).

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy that involves taking white blood cells from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient. These cells are called Tumor Infiltrating Lymphocytes, or TIL and we have given this type of treatment to over 100 patients. In this study, we are selecting a specific subset of white blood cells from the tumor that we think are the most effective in fighting tumors and will use only these cells in making the tumor fighting cells.

Objective:

The purpose of this study is to see if these specifically selected tumor fighting cells can cause melanoma tumors to shrink and to see if this treatment is safe.

Eligibility:

- Adults age 18-70 with metastatic melanoma who have a tumor that can be safely removed.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Surgery: If the patients meet all of the requirements for the study they will undergo surgery to remove a tumor that can be used to grow the TIL product.
* Leukapheresis: Patients may undergo leukapheresis to obtain additional white blood cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the tumor infiltrating lymphocytes (TIL) cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

...

DETAILED DESCRIPTION:
Background:

* Autologous tumor infiltrating lymphocytes (TIL) followed by high dose aldesleukin can mediate the regression of bulky metastatic melanoma when administered to a patient following a non-myeloablative but lymphodepleting chemotherapy preparative regimen.
* In animal models, mixing irrelevant (non-reactive) cells with tumor-reactive cells negatively impacts on tumor treatment possibly by competing for cytokines, suggesting that enrichment for tumor-reactive cells could enhance clinical efficacy. Additionally, preclinical animal models and clinical investigation have demonstrated that prolonged in vitro culture negatively impacts on tumor treatment.
* The current method for enrichment of tumor-reactive TIL requires screening of multiple independent TIL cultures for anti-tumor specificity using gamma-interferon production by TIL. However, in vitro screening depends on autologous tumor reagents that are often unavailable, and interferon (IFN) gamma release in vitro may not be the best effector function to evaluate tumor recognition. The screen increases the length of in vitro culture times (30 days), which results in shorter telomere lengths and more differentiated cells. Additionally, selection of a few highly reactive cultures for further expansion may reduce the diversity of cluster of differentiation 8 (CD8+) repertoire recognizing the tumor.
* 4-1BB is a co-stimulatory molecule up-regulated on the cell surface of T cells upon T-cell receptor (TCR) engagement. Pre-clinical studies in the Surgery Branch have evaluated a fast and simplified method to select and expand a diverse tumor-reactive repertoire, regardless of knowledge of the specific antigen recognized, based on selection of 4-1BB expressing TIL from the fresh tumor digest.

Objectives:

* To determine the safety and objective response rate of patients with metastatic melanoma receiving ACT using 4-1BB selected TIL plus aldesleukin treatment following a chemotherapy preparative regimen.
* To determine the survival of patients receiving this treatment regimen.

Eligibility:

Patients who are 18 years or older must have:

* Evaluable metastatic melanoma;
* Metastatic melanoma lesion suitable for surgical resection for the preparation of TIL;
* No contraindications to high-dose aldesleukin administration;
* No concurrent major medical illnesses or any form of immunodeficiency

Design:

* Patients with metastatic melanoma will have a lesion resected and 4-1BB expressing tumor infiltrating lymphocytes will be isolated using a fluorescence-activated cell sorting (FACS) sorter approved for clinical use. The 4-1BB selected cells will be rapidly expanded in vitro and administered plus aldesleukin following a non-myeloablative chemotherapy preparative regimen.
* The study will be conducted using a stage 2 optimal design to determine if this treatment is able to be associated with a clinical response rate that can rule out 10% (p0=0.10) in favor of a modest 30% partial response (PR) + complete response (CR) rate (p1=0.30).
* Up to 35 patients may be enrolled over 2 years.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma with at least one lesion that is resectable for tumor infiltrating lymphocytes (TIL) generation. The lesion must be at least 1 cm in diameter that can be surgically removed with minimal morbidity (defined as any operation for which expected hospitalization <less than or equal to days).
2. Confirmation of diagnosis of metastatic melanoma by the Laboratory of Pathology of the National Cancer Institute (NCI).
3. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible.
4. Greater than or equal to 18 years of age and less than or equal to age 70.
5. Able to understand and sign the Informed Consent Document
6. Willing to sign a durable power of attorney
7. Clinical performance status of Easter Cooperative Oncology Group (ECOG) 0 or 1
8. Oxygen saturation of greater than or equal to 90% on room air
9. Life expectancy of greater than three months
10. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
11. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
12. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
13. Hematology

    * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim
    * White blood cell (WBC) greater than or equal to 3000/mm^3
    * Platelet count greater than or equal to 100,000/mm^3
    * Hemoglobin > 8.0 g/dl
14. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal
    * Serum creatinine less than or equal to 1.6 mg/dl
    * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dl.
15. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients must have progressing disease after prior treatment.

    Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in Section 2.1.1.
16. Six weeks must have elapsed from the time of any antibody therapy that could affect an anti cancer immune response, including anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4) antibody therapy at the time the patient receives the preparative regimen to allow antibody levels to decline.

Note: Patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Prior treatment with an anti-4-1BB antibody.
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
3. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
6. Concurrent systemic steroid therapy.
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization or ischemic symptoms.
9. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45%, testing is required in patients with:

   * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   * Age greater than or equal to 60 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Atkins MB, Kunkel L, Sznol M, Rosenberg SA. High-dose recombinant interleukin-2 therapy in patients with metastatic melanoma: long-term survival update. Cancer J Sci Am. 2000 Feb;6 Suppl 1:S11-4. PMID 10685652
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lymphocyte Depleting Prep Regimen
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lymphocyte Depleting Prep Regimen
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v3.0. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 2 years and 59 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphocyte Depleting Prep Regimen
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Objective Response Rate of Patients With Metastatic Melanoma
Description: Objective response is defined as complete response + partial response and was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: approximately 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Lymphocyte Depleting Prep Regimen
Number analyzed (Participants) | 6
percentage of participants
  Progressive Disease | 83.33
  Partial Response | 16.67
  Complete Response | 0
  Stable Disease | 0

3. Secondary Outcome: Overall Survival (OS) of Patients Receiving a Lymphocyte Depleting Preparative Regimen
Description: OS is defined as the time between the first day of treatment to the day of death or date last known alive.
Time Frame: up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Lymphocyte Depleting Prep Regimen
Number analyzed (Participants) | 6
months | 12 [2 to 35]

ADVERSE EVENTS:
Time Frame: 2 years and 59 days
Arm/Group | Lymphocyte Depleting Prep Regimen
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphocyte Depleting Prep Regimen (N=6)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 6 (6)
Platelets (Blood and lymphatic system disorders) | 6 (6)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No